# Wise Interventions for Adolescents and Young People in the Digital Society

# **University of Deusto**

PR[18]\_SOC\_0096 (BBVA foundation)

**Informed Consent Form** 

May 31, 2020

# Faculty of Psychology and Education University of Deusto

This consent form provides information on a research project that is being carried out at your child's school in collaboration with the University of Deusto and that aims to evaluate the effectiveness of short wise interventions to improve the quality of adolescents' and young people's social relations the digital society.

Below you will find all the relevant information about the project. After you have read the information, if you do **not** want your child to participate in this project, please fill out the consent form and return it to your child's school **in 3 days**. If you authorize your child to participate, you **do not have to complete the form or return it**.

### 1. Purpose of the project:

The objective of this project is to implement various intervention formats to determine which of them is the most effective. The interventions aim to enhance prosocial behaviors such as empathy, generosity, and solidarity on the Internet, while seeking to reduce online risks such as bullying and other phenomena that threaten young people.

The intervention takes place in a single session of about 50 - 60 minutes. We employ two intervention formats to which the participants are randomly assigned. Afterwards, everyone will have the opportunity to receive the intervention that is the most effective.

The intervention consists of exercises such as: (1) reading scientific information about social behavior and its role in the well-being of individuals, (2) self-affirmation of positive values, (3) reading, reflecting, and writing about the meaning and value of prosocial behaviors and online risk behaviors through stories and their own experiences and those of other young people of their age.

All the students in your child's class have received the invitation to participate.

### 2. What will my child be asked to do?

If you allow your child to participate in this study, he/she will be asked to:

- Participate in the 50-minute intervention.
- Complete a questionnaire of about 30-40 minutes one week before and three and six months after the intervention.

# 3. How will the researchers protect the participants' privacy?

The study was funded by the BBVA Foundation and with the approval of the Committee of Ethics in Research at the University of Deusto. The researchers will protect the privacy of all the participants. No names or surnames are indicated in any place. The evaluation and intervention data will be joined by a code only known to the participant.

# 4. How will the researchers share the results of the project?

Your child's school will receive a preliminary and final report which will reflect the results of the evaluation of the program and will be distributed to all the parents.

# 5. Is there any risk or benefit for my child?

There are no foreseeable risks associated with participation in this project. The intervention and the questionnaires are regular school activities. The intervention can be beneficial for a high percentage of students.

# 6. Does my child have to participate?

Consent is optional. Your decision to allow or forbid your child to participate will not affect your child's current or future relationship with the University of Deusto, the school, or the teacher. If you choose to allow your child to participate, he/she will be asked if he/she agrees to participate, and if your child to accepts, he/she will receive all necessary instructions. In addition, he/she is free to stop participating at any time without any penalty or adverse consequence. You can also initially allow your child to participate in the study and then change your mind without any kind of penalty.

This research study will take place during the normal classroom activities. However, if you do not want your child to participate, there will be a different activity available for him or her. Your child will be offered the possibility to use the time to read or do homework.

#### 7. What will happen if my child does not want to participate?

In addition to your permission, your child must agree to participate in the study. If he or she does not wish to participate, he/she will not be included in the study, and no there will be no penalty. Even if he/she initially agreed to participate in the study, he/she can change his/her mind later on without any penalty.

# 8. Is there any compensation?

There will be no compensation for participating. However, gift vouchers will be drawn to exchange in a department store in each classroom among the participants.

# 9. Who has reviewed the study?

This research study has been approved and funded by "BBVA Foundation Grants to Scientific Research Teams in the areas of Economics and Digital Society; Digital Humanities; Big Data; Biomedicine; Ecology and Conservation Biology" in the 2018 call. The project has also been reviewed by the Ethics Committee of the University of Deusto and by the directors of the schools. The school will not carry out the project activities. The study will be carried out by researchers from the University of Deusto.

# 10. Who can I contact if I have questions about the study?

Before, during, or after your participation, you can contact any of the following people:

[masked]

| Your signature indicates that you have read the information and have decided not to allow your child to participate in this project. If you give your permission for your child to participate, you need not complete this form. NO, my son/daughter may NOT participate in the project. | |
|---|---|
| Name and surname of the Student | |
| Signature of the Father/Mother or Guardian | Date |

The form must only be signed if you **do not** want your child to participate